CLINICAL TRIAL: NCT03760835
Title: Congenital Adrenal Hyperplasia: Innovative Once Daily Dual Release Hydrocortisone Treatment
Brief Title: Congenital Adrenal Hyperplasia Once Daily Hydrocortisone Treatment
Acronym: CareOnTIME
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof. Rosario Pivonello, Full Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140/16
Record Dates: First submitted 2018-11-09; First posted 2018-11-30 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: congenital adrenal hyperplasia; glucocorticoid treatment; dual release hydrocortisone
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Cortisone; Prednisone; Prednisolone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual-release hydrocortisone (Experimental)
  Interventions: Drug: Conventional Glucocorticoids (immediate release hydrocortisone, cortisone acetate, prednisone, prednisolone, dexamethasone); Drug: Dual release hydrocortisone (plenadren)
- Conventional glucocorticoids (Active Comparator)
  Interventions: Drug: Conventional Glucocorticoids (immediate release hydrocortisone, cortisone acetate, prednisone, prednisolone, dexamethasone)

INTERVENTIONS:
Drug: Conventional Glucocorticoids (immediate release hydrocortisone, cortisone acetate, prednisone, prednisolone, dexamethasone) — Treatment of congenital adrenal hyperplasia
Drug: Dual release hydrocortisone (plenadren) — Treatment of congenital adrenal hyperplasia
  Arms: Dual-release hydrocortisone

SUMMARY:
This is a controlled, open study designed to compare the effects of dual-release hydrocortisone preparations versus conventional glucocorticoid therapy on clinical, anthropometric parameters, metabolic syndrome, hormonal profile, bone status, quality of life, reproductive, sexual and psychological functions and treatment compliance in patients affected by congenital adrenal hyperplasia due to 21 OH deficiency.

DETAILED DESCRIPTION:
Congenital adrenal hyperplasia due to 21-hydroxylase deficiency is an autosomal recessive disorder characterized by cortisol and in some cases aldosterone deficiency, associated with androgen excess. Treatment goals are to replace cortisol deficiency, to control androgen levels, while avoiding the adverse effects of exogenous glucocorticoids. A variety of glucocorticoid treatments have been used in an attempt to control the overnight increase in adrenal androgens. However, there is no consensus on the optimum management of congenital adrenal hyperplasia adults. Current evidence in patients with adrenal insufficiency suggests that the inability of current regimens to replace physiological circadian cortisol levels, leads to adverse clinical outcomes, including metabolic syndrome, insulin resistance, increased risk factors for cardiovascular diseases, bone and immune alterations, sleep disturbances and quality of life impairment. Moreover, the risk for poor treatment compliance, in case of multiple daily doses treatment regimens, should not be excluded. In this trial a dual-release hydrocortisone preparation, that been able to mimic the circadian pattern of circulating cortisol, was studied in patients with adrenal insufficiency due to congenital adrenal hyperplasia.

All patients with a diagnosis of congenital adrenal hyperplasia due to 21-hydroxylase deficiency, irrespective of glucocorticoid treatment, are eligible for the inclusion in the study and may be asked to participate in the study. Patients are followed during the course of routine clinical practice for the duration of time that the study is active.

ARM1: Conventional glucocorticoid therapy is continued as before entering the study

ARM2: Dual release hydrocortisone oral tablets is administered once-daily in the fasting state. The dose is kept the same as patients had before entering the trial.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged >18 years;
* established diagnosis of adrenal insufficiency in congenital adrenal hyperplasia due to 21-hydroxylase deficiency;
* stably treated with conventional glucocorticoids, available to change their regimen according to random allocation
* written informed consent/assent to participate in the study in compliance with local regulations.

Exclusion Criteria:

* clinical or laboratory signs of severe cerebral, respiratory, hepatobiliary or pancreatic diseases, renal dysfunction, gastrointestinal emptying, or motility disturbances (i.e. chronic diarrhea), significant psychiatric illnesses;
* history of/or current alcohol and/or drug abuse;
* night shift workers;
* underlying diseases that could necessitate treatment with glucocorticoids;
* therapies with hepatic enzyme induction drugs interfering with glucocorticoid kinetics, or immunosuppressive steroid therapy;
* patients with a documented intolerance/known hypersensitivity to dual release hydrocortisone;
* vulnerable populations, such as elderly, cancer patients, pregnant and lactating women;
* history of non-compliance to medical regimens, or potentially unreliable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-08-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in measurement of total and LDL cholesterol (mg/dl) | 0, + 6 months, + 12 months, +24 months
  Single outcome measurement of cholesterol levels (mg/dl)

SECONDARY OUTCOMES:
Change from baseline in measurement of glycaemia (mg/dl) | 0, + 6 months, + 12 months, +24 months
  Measure of glycaemia (mg/dl)
Change from baseline in measurement of BMI (Kg/m2) | 0, + 6 months, + 12 months, +24 months
  Measure of BMI (Kg/m2)
Change from baseline in measurement of blood pressure (mmHg) | 0, + 6 months, + 12 months, +24 months
  Measure of blood pressure (mmHg)
Change from baseline in measurement of insulinemia (μU/mL) | 0, + 6 months, + 12 months, +24 months
  Measure of insulinemia (μU/mL)
Change from baseline in measurement of triglycerides (mg/dl) | 0, + 6 months, + 12 months, +24 months
  Measure of triglycerides (mg/dl)
Change from baseline in measurement of HDL-cholesterol (mg/dl) | 0, + 6 months, + 12 months, +24 months
  Measure of HDL-cholesterol (mg/dl)
Change from baseline in measurement of Glycated Haemoglobin (%) | 0, + 6 months, + 12 months, +24 months
  Measure of Glycated Haemoglobin (%)
Changes in bone mineral density | 0, + 12 months, +24 months
  Bone mineral density quantified by Dual X-Ray Absorptiometry (DEXA)]
Changes in quality of life | 0, + 6 months, + 12 months, +24 months
  Quality of life will be measured by Addison Quality of Life (AddiQol) questionnaire, used to assess quality of life in patients suffering from adrenal insufficiency. Each question has a score ranging from 1 to 4. Total score (minimum: 30; maximum: 120) is obtained summing each question score. The higher the scores are, the better the quality of life is. No clear cut-offs are defined.
Changes in sex function in males | 0, + 6 months, + 12 months, +24 months
  Sex function will be measured by International Index of Erectile Function (IIEF) questionnaire. IIEF is divided into five function domains: Erectile function (Q1-5, Q15; score range Q1-5: 0-5; score range Q15: 1-5), Orgasmic function (Q9-10; score range Q9: 0-5; score range Q10: 1-5), Sexual desire (Q11-12; score range: 1-5), Intercourse satisfaction (Q6-8; score range: 0-5), Overall satisfaction (Q13-14; score range: 1-5). The higher the domain scores are, the better the male sexual functions are.
Changes in sex function in females | 0, + 6 months, + 12 months, +24 months
  Sex function will be measured by Female Sexual Function Index (FSFI) questionnaire. FSFI is divided into six domains: Desire (Q1-2; score range: 1-5), Arousal (Q3-6; score range: 0-5), Lubrification (Q7-10; score range: 0-5), Orgasm (Q11-13; score range: 0-5), Satisfaction (Q14-16; score range Q14: 0-5; score range Q15-16: 1-5), Pain (Q17-19; score range: 0-5). To obtain the full scale score (ranging from 2 to 36), each domain score range should be corrected by an individual factor (Desire: 0.6; Arousal and Lubrification: 0.3; Orgasm, Satisfaction and Pain: 0.4). The higher the score is, the better the female sexual function is.
Changes in depression status | 0, + 6 months, + 12 months, +24 months
  Depression status will be measured by Beck Depression Inventory Test (BDI-II) questionnaire. Each question has a score ranging from 0 to 3. Total score (minimum: 0; maximum: 63) is obtained summing each question score. Scores range from minimum (0-13), mild (14-19), moderate (20-28), severe (29-63)
Incidence of Treatment Adverse Events (safety analysis) | 0, + 6 months, + 12 months, +24 months
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 4.0 (not a scale)
Changes in androgens levels | 0, + 6 months, + 12 months, +24 months
  Measure of androstenedione/testosterone ratio
Changes in sperm concentration | 0, + 6 months, + 12 months, +24 months
  Evaluation of sperm concentration according to WHO criteria
Changes in ovarian follicles reserve | 0, + 6 months, + 12 months, +24 months
  Evaluation of number of ovarian follicles by conventional ultrasound imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University, Naples, Italy

IPD SHARING:
Plan to Share IPD: No